CLINICAL TRIAL: NCT00929500
Title: The Effect of Mixed Aerobic and Strength Training Program on Physical Fitness and Cerebrovascular Function in Older Women With Metabolic Syndrome: A Pilot Study With Randomized Control Trial (RCT) Design
Brief Title: Exercise Program in Women With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Vera Novak, Associate Professor of Neurology, Director Safe Laboratory, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2009P000121
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MAST program (Experimental): Mixed Aerobic and Strength Training program (MAST): Each exercise session consisted of 10 minutes of warm-up, 15-30 minutes of interval aerobic training by cycle ergometer according to the program, 20 minutes of strength training exercises, and 10 minutes of cool-down by stretching.
  Interventions: Behavioral: MAST program
- UC (No Intervention): Usual Care (UC) with Educational Lectures: No exercise sessions.

INTERVENTIONS:
Behavioral: MAST program — MAST program: twice a week for 4 months
  Arms: MAST program

SUMMARY:
The purpose of this study is to test whether a supervised mixed aerobic and strength training (MAST) program is effective in improving overall physical fitness and blood flow in the brain and lowering risk factors of coronary artery disease (CAD) in women with metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome is a cluster of conditions and disorders that increase the risk for coronary artery disease (CAD) and strokes. Sedentary lifestyle is one of the risk factors, which decrease overall physical fitness and together with aging may lead to decrease in physical functioning in everyday life as well as changes in blood flow in the brain and cognitive functions. Regular physical activity is associated with a reduced risk of cardiovascular disease. It may also improve blood flow velocity and cognitive functions. Physical activity should be as effective as possible, but also as safe as possible. Supervised mixed aerobic and strength training (MAST) program for 4 months enables to individualize the intensity of aerobic exercise based on measured maximal exercise capacity. Throughout each training session heart rate will be monitored with a new real time wireless ECG system.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Age 50 or over
* Diagnosed metabolic syndrome

Exclusion Criteria:

* Any unstable or acute medical condition that the study physician deem unsafe for participation
* Positive stress test for CAD or other ischemic conditions
* Myocardial infarction or major surgery within 6 months
* History of a clinically documented stroke
* Clinical dementia (by history) or inability to follow details of the protocol
* Carotid stenosis > 50% by medical history
* Insulin dependent diabetes mellitus (also type II, if using insulin) or history of severe hypoglycemic episodes within 6 months requiring hospitalization
* Liver or renal failure or transplant
* Severe blood pressure elevation (systolic BP > 180 and/or diastolic BP > 110 mm Hg)
* Anemia (Hb < 10)
* Seizure disorders
* Current recreational drug or alcohol abuse
* BMI > 45, but body weight under 280 lbs
* Inability to obtain permission for participation from the primary care physician
* Clinically significant and movement limiting hip, knee and/or back disorders or injury, and rheumatoid arthritis
* Transcranial Doppler (TCD) exclusion criteria - poor insonation window and TCD signal

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Novak, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Harvard University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heli V, Ihab H, Kun H, Brad M, Jessica W, Vera N. Effects of exercise program on physiological functions in postmenopausal women with metabolic syndrome. Int J Gerontol. 2013 Dec;7(4):231-235. doi: 10.1016/j.ijge.2013.05.002. PMID 24634702

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 subjects were consented. Of those, 16 were determined ineligible to participate. 12 subjects were randomized (8 to intervention group and 4 to control group). At the end of the trial, only 4 intervention and 4 sontrol subjects completed the study.
Groups:
- MAST Program: Mixed Aerobic and Strength Training program (MAST)
  MAST program: MAST program: twice a week for 4 months
- Usual Care: Usual Care (UC) with Educational Lectures
Period: Overall Study
Arm/Group | MAST Program | Usual Care
Started | 8 | 4
Completed | 4 | 4
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAST Program | Usual Care | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.25 (8.9) | 55.75 (6.07) | 58 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximal Oxygen Uptake
Description: To obtain peak oxygen uptake (VO2max; ml-1/min-1/kg), a symptom-limited exercise stress test was performed on a cycle ergometer. The test was preceded by a 2-minute warm-up at the intensity of 20 W. The first test load was 20 W, and was increased by 20 W at each 2-minute stage until the participants could no longer continue, i.e., they were unable to maintain pedaling frequency > 40 rpm, they achieved a respiratory exchange ratio of more than 1.0, or clinical criteria for test termination was observed. VO2max was measured and monitored with a breath-by-breath gas exchange system.
Time Frame: At baseline and after 4 months of intervention
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | MAST Program | Usual Care
Number analyzed (Participants) | 4 | 4
ml/kg/min
  Baseline | 18.3 (3.8) | 15.8 (5.0)
  Week 16 | 18.6 (3.7) | 14.4 (4.4)

2. Secondary Outcome: Cerebral Blood Flow Velocity (BFV)
Description: Cerebral BFV was monitored using Transcranial Doppler Ultrasound.11 The middle cerebral artery was insonated from the temporal window by placing the 2-MegaHertZ (MHz) probe against the skin of the temporal region above the zygomatic arch. The probe was positioned to obtain maximal BFV and was fixed at the desired angle using a 3-dimensional positioning system. Once instrumented, BFV was continuously recorded throughout ten minutes of supine rest and 10-minutes on a table tilted to 80° from the horizontal position (head-up with foot plate support).
Time Frame: At baseline and after 4 months of intervention
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | MAST Program | Usual Care
Number analyzed (Participants) | 4 | 4
cm/s
  Baseline (supine) | 37.4 (11.7) | 41.7 (31.9)
  Week 16 (supine) | 34.7 (15.8) | 33.9 (15.7)
  Baseline (standing) | 33.3 (7.4) | 36.7 (26.3)
  Week 16 (standing) | 33.2 (16) | 37.8 (5.4)

3. Secondary Outcome: Trail Making Test
Description: The Trail Making (TM) test is a measure of shifting attention. Participants are required to sequentially connect a series of numbered circles (Part A), and then to alternate between numbers and letters sequentially (Part B) (e.g., A-1-B-2-C-3..). Any participant who has not completed Part B within the standard 5 minutes (300 seconds) allotted for the task will be considered unable to complete the task. The scores in Part A (TM-A), Part B (TM-B) T scores ( age, education adjusted), and their difference (TM-B -TM-A) were calculated and used to measure executive function, i.e., lower scores indicates better performance.
Time Frame: At baseline and after 4 months of intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MAST Program | Usual Care
Number analyzed (Participants) | 4 | 4
T-score
  Trail Making A (Baseline) | 29.1 (10.9) | 31.2 (9.3)
  Trail Making B (Baseline) | 78.4 (22.7) | 64.9 (31.8)
  Trail Making B-A (Baseline) | 49.3 (19.2) | 33.7 (22.9)
  Trail Making A (Week 16) | 24.9 (7.7) | 29.7 (15.9)
  Trail Making B (Week 16) | 65.6 (23) | 59.8 (14.8)
  Trail Making B-A (Week 16) | 40.8 (21.2) | 30.2 (2.6)

4. Secondary Outcome: Muscle Strength
Description: MAST sessions were held twice a week for 16 weeks. Each exercise session consisted of 10 min of warm-up, 15-30 min of interval aerobic training by cycle ergometer according to the program, 20 min of strength training exercises, and 10 min of cool-down by stretching. The target heart rate (HR) increased progressively from 50% up to 80% of HR reserve by the end of the intervention period.The Karvonen formula ([(HRmax - HRrest)×(0.50 to 0.80)] + HRrest) was used to calculate the target HR. During every training session a new wireless computerized ECG monitoring system was used. After aerobic training, the strength training program was performed. Exercises used body mass as resistance and included squat, step-up-squat, step-up, heel rise, and sit-ups. Dumbbells were used as extra weight (5 or 10% of body weight) during other exercises except for sit-ups. The control group participated in an educational session once a month and kept physical activity diaries during the intervention period.
Time Frame: At baseline and after 4 months of intervention
Measure: Mean (Standard Deviation); unit: W
Arm/Group | MAST Program | Usual Care
Number analyzed (Participants) | 4 | 4
W
  Baseline | 96.7 (19.7) | 95 (19.1)
  Week 16 | 103.3 (23.4) | 90 (25.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MAST Program | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAST Program (N=8) | Usual Care (N=4)
Myocardial infarction (Cardiac disorders) | 1 | 0 — Subject suffered a myocardial infarction during a gastric bypass surgery after enrollment in study and randomized, but prior to starting the exercise training program.

LIMITATIONS AND CAVEATS:
Difficulty in recruiting older women with Metabolic syndrome, unwilling to participate due to time commitment and transportation difficulties, interrupt the recruitment process due to time constraints. Results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No